CLINICAL TRIAL: NCT05980884
Title: Evaluation of Microbial-derived TMAO Production From Carnitine Intake by Testing Fecal Gbu Gene
Brief Title: Using Gut Microbial Gbu Gene Testing to Estimate Host TMAO Production Capacity
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 202303144RINA
Record Dates: First submitted 2023-07-20; First posted 2023-08-08 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Gut Dysbiosis for TMAO Production From L-carnitine Consumption
Keywords: gbu gene cluster; TMAO; gut microbiota; red meat; cardiovascular disease
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Carnitine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- L-Carnitine supplementation (Experimental): Participants are required to take a capsule containing 500mg L-carnitine/day continuous for 7-10 days. During the intervention, participants are asked to collect urine sample and dietary record each day. Blood and fecal samples will be collected before and after the intervention. Each participant needs to complete a food frequency questionnaire.
  Interventions: Dietary Supplement: L-carnitine

INTERVENTIONS:
Dietary Supplement: L-carnitine — Participants are required to take a capsule containing 500mg L-carnitine/day continuous for 7-10 days.

SUMMARY:
The risk of cardiovascular diseases from red meat consumption varies among individuals due to variations in gut microbiota. L-carnitine in red meat can be converted to TMAO in the body by certain bacteria. Not everyone experiences a significant increase in TMAO levels after consuming carnitine. Gut microbiota differences are observed between high and low TMAO producers. The presence of the gbu gene in gut microbiota is linked to TMAO production. This clinical research aims to determine if the gbu gene can predict TMAO levels after dietary carnitine intake.

DETAILED DESCRIPTION:
The risk of developing cardiovascular diseases due to the consumption of red meat varies among individuals, and this may be attributed to differences in the composition and function of gut microbiota. Studies have found that red meat, rich in L-carnitine, may be metabolized by certain anaerobic bacteria in the intestines to produce trimethylamine N-oxide (TMAO) in the human body. Previous research utilizing the oral carnitine challenge test (OCCT) revealed that not everyone experiences a significant increase in blood TMAO levels after consuming carnitine. Moreover, individuals with high TMAO production and low TMAO production showed distinct differences in their gut microbiota.

Furthermore, we have discovered a significant correlation between the abundance of the gbu gene in gut microbiota and the production of TMAO in response to dietary carnitine intake. Therefore, through the design of clinical research, we aim to investigate and assess whether the abundance of the gbu gene in gut microbiota can predict the levels of TMAO produced in the human body under dietary carnitine intake.

ELIGIBILITY:
Inclusion Criteria:

* Adult with age between 18 to 70
* Must be able to swallow tablets

Exclusion Criteria:

* Antibiotics use within one month
* L-carnitine supplement use within one month
* Chronic diarrhea
* Myasthenia gravis
* Diabetes mellitus
* Parathyroid disorders
* Chronic kidney disease
* Epilepsy
* Severe anemia
* Cardiovascular diseases.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2023-07-24 (Actual); Primary Completion 2026-04-25 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Blood TMAO level measured by LC-MS/MS | up to 7-10 days
Urine TMAO level measured by LC-MS/MS | up to 7-10 days
Fecal gbuB gene abundance measured by qPCR | up to 7-10 days

SECONDARY OUTCOMES:
Carnitine intake measured by 24hr dietary record | up to 7-10 days
Gut microbiome profiles measured by shotgun metagenome sequencing | up to 7-10 days

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
The data will be uploaded to be public when the research is published

REFERENCES:
- [Result] Wu WK, Lo YL, Chiu JY, Hsu CL, Lo IH, Panyod S, Liao YC, Chiu THT, Yang YT, Kuo HC, Zou HB, Chen YH, Chuang HL, Yen JJY, Wang JT, Chiu HM, Hsu CC, Kuo CH, Sheen LY, Kao HL, Wu MS. Gut microbes with the gbu genes determine TMAO production from L-carnitine intake and serve as a biomarker for precision nutrition. Gut Microbes. 2025 Dec;17(1):2446374. doi: 10.1080/19490976.2024.2446374. Epub 2024 Dec 26. PMID 39722590